CLINICAL TRIAL: NCT00436995
Title: A Multicentre, Single Arm Study Evaluating The Extension From Weekly To Once Every Other Week Darbepoetin Alfa Administration In Subjects With Chronic Kidney Disease Receiving Dialysis.
Brief Title: Extension From Weekly to Once Every Other Week Darbepoetin Alfa Administration in Subjects With Chronic Kidney Disease Receiving Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20050210
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Last update posted 2011-01-21 (Estimated); Status verified 2011-01

CONDITIONS: Chronic Kidney Disease
Keywords: Dialysis; Anaemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia | interventions — Darbepoetin alfa

ARMS (1):
- Single (Other)
  Interventions: Drug: Darbepoetin Alfa

INTERVENTIONS:
Drug: Darbepoetin Alfa — Administered IV or SC, Q2W at the following unit doses: 10, 15, 20, 30, 40, 50, 60, 80, 100, 130, 150, 200 or 300ug. Initial Q2W dose calculated from pre-enrollment QW doses. Doses titrated to achieve target Hb.

SUMMARY:
The purpose of this study is to assess the proportion of subjects sucessfully achieving a mean Hemoglobin greater than or equal to 11 g/dL during the evaluation period following extension from Weekly (QW) to Once Every Other Week (Q2W) Darbepoetin Alfa administraion.

ELIGIBILITY:
Inclusion Criteria:

* Receiving dialysis for 3 months or more before enrollment.
* The mean of 2 screening Hb values taken at least 7 days appart must be greater than or equal to 11g/dL and less than or equal to 13.0 g/dL
* Receiving stable QW darbepoetin alfa doses for at least 6 weeks before enrollment
* Adequate iron stores (serum ferritin equal to or greater than 100 ug/L

Exclusion Criteria:

* Uncontrolled hypertension
* Prior history of Cardiovascular Incidents 12 weeks prior to enrollment
* Other hematological disorders
* Upper or lower GI bleed within the prior 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2006-04; Primary Completion 2007-01 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Haemoglobin values to be maintained at greater than 11.0 g/dL during the evaluation period. | 33 weeks

SECONDARY OUTCOMES:
Q2W doses over duration of study. | 33 weeks
Hb values during the evaluation period. | 33 weeks
adverse events during study | 33 weeks
Hb Rate of Rise during study and excursions above 14g/dL | 33 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com